CLINICAL TRIAL: NCT04851431
Title: Effects of Peer Mentoring on Caregivers of Patients With Acquired Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Michael Jones, Director Emeritus, Virginia C Crawford Research Institute, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1543747
Record Dates: First submitted 2021-04-08; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Acquired Brain Injury; Family Members
Keywords: Peer-to-peer mentoring in self management; Acquired Brain Injury; Family Caregivers; Caregiver stress and burden
MeSH Terms: conditions — Brain Injuries; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-to-One Peer Mentoring (Experimental): Caregiver will be matched based on characteristics such as age, date of patient injury, level of patient injury, cause of patient injury, marital status, work status before and after patient injury, interests, and leisure activities. After participant is matched with a peer mentor, they will be required to have at least one weekly one-to-one interaction from time of match until 30 days post- discharge.
  Interventions: Behavioral: one-to-one peer mentoring
- Usual Care (Active Comparator): Participants received the usual discharge planning and family support services offered by the ABI program. These services include nurse instruction in care routines, case management support for discharge, peer support services, referral to family counseling and community services as indicated, and general information resources about brain injury. Participants in both the intervention and usual care groups also had access to the online peer support community created for ABI caregivers (facebook.com/shepherdbi.peers). In addition, usual care participants could request one-to-one visits with peer mentors and, indeed, most usual care participants received at least one peer mentoring visit.
  Interventions: Behavioral: one-to-one peer mentoring

INTERVENTIONS:
Behavioral: one-to-one peer mentoring — Weekly meetings with a peer family caregiver

SUMMARY:
Family caregivers often take on the demands of long-term caregiving after ABI. Early efforts to prepare family caregivers for the caregiving role after discharge from acute ABI inpatient rehabilitation may be beneficial in many ways. This study will look at the impact of participation in a one-to-one peer mentor program on the use of family support services and caregivers' emotional health and well-being (depression symptoms, stress).

Participants in this study will include caregivers of patient admitted to the Shepherd Center ABI inpatient rehabilitation unit. Caregivers will be randomly selected to participate in the one-to-one mentor program. The program will include visits with a peer mentor who is the caregiver of an individual with an acquired brain injury. Participants will be able to choose a peer mentor that matches their personal situation and preferences. They will meet with the peer mentor about once a week during the patient's stay at Shepherd Center and may continue with phone calls up to 30 days post-discharge. Participants will be asked to complete a brief evaluation after each peer mentor interaction to determine the value of the interactions and their interest in continuing visits. Participants will be asked to take part in three interviews that will last 10-15 minutes. The first will be within the first two weeks at Shepherd Center and the second will be a few days after discharge. A third interview will be conducted by phone about 30 days post discharge.

DETAILED DESCRIPTION:
The one-to-one peer mentor intervention will be evaluated for effectiveness on caregiver outcomes and use of family support services. 40 participants will be enrolled to assess the impact of one-on-one peer mentor relationships through the completion of the Kingston Caregiver Stress Scale (KCSS), Patient Health Questionnaire (PHQ-9), and participation in family support classes.

Participants will be recruited, based on inclusion and exclusion criteria, via in person meeting, by the study's research coordinator at Shepherd Center. Once a recruited subject expresses interest in participating in the study, the research coordinator will go over the informed consent form with the participant and enroll them into the study.

Once informed consent is obtained, enrolled participants will be asked to answer questions about their demographics and psychological well-being (PHQ-9 and KCSS). At this time, the participant will be randomized into the peer mentor intervention group or the control group (receiving general peer support under usual care).

1. Usual Care Peer Support Family support services offered at Shepherd Center under usual care involves peer mentoring, community support, brain injury education classes, and workshops. Within 5-10 days of admission, the caregiver of the patient is introduced to the peer support team. Caregivers are seen by peer mentors within the family support services on a referral basis from therapists, nurses, counselors, or physicians or on request from the caregivers/family. There are no scheduled interactions between peer support and the caregiver, nor is the caregiver assigned a peer mentor. The family is made aware of resources, but participation is optional for the family/caregiver. Access to the ABI Peer Support Facebook page is also available and the page is maintained by the Shepherd Peer Mentors.
2. One-to-One Mentoring Caregiver will be matched based on characteristics such as age, date of patient injury, level of patient injury, cause of patient injury, marital status, work status before and after patient injury, interests, and leisure activities. After participant is matched with a peer mentor, they will be required to have at least one weekly one-to-one interaction from time of match until 30 days post- discharge. The use of family support services by the participant will be monitored by peer mentor reported interactions, as well as attendance in family support classes. The participant will be asked to briefly review each weekly scheduled one-to-one interaction to ensure mentorship needs are being met on behalf of the participant.

Participant use of family support services offered by Shepherd Center will be monitored by attendance and by self-reported use of resources by caregiver, to peer mentors. Peer support documentation is recorded after each interaction by the peer mentor. Information logged includes the date, duration of interaction, type of interaction, and topics discussed. Attempts made at communicating with caregiver is also documented by the peer mentor within the database. C

Before discharge from Shepherd Center, the participant will be asked to answer questions about their medical history, family history, and psychological well-being. At 30 days post discharge, participants will be asked to answer questions about their psychological well-being (PHQ-9, KCSS). Those in the intervention group will also be asked to give feedback on the one-to-one peer mentor program (One-to-one Peer Mentor Initiative Survey).

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for rehabilitation off acquired brain injury Planned discharge to home Family caregiver aged 18 years or older English-speaking

Exclusion Criteria:

* Discharge location is not home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Participation in family support services | Attendance documented for all classes and meetings held during patients' inpatient stay; average inpatient length of stay is 52 days
  Number of peer support meetings, family orientation classes, and caregiver self-management classes attended by family caregivers during the inpatient stay.
Change in Kingston Caregiver Stress Scale (KCSS) scores | 1) baseline, at time of enrollment in the study; 2) within 72 hours of discharge to home; 3) 30-days post-discharge
  Caregiver stress and burden; scores range from 10-50; higher score reflects higher stress
Change in Patient Health Questionnaire - 9 (PHQ-9) scores | 1) baseline, at time of enrollment in the study; 2) within 72 hours of discharge to home; 3) 30-days post-discharge
  Caregiver depressive symptoms; scores range from 0-27; higher score reflects higher depression

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No